CLINICAL TRIAL: NCT01608399
Title: A Randomized Controlled Trial of the Effectiveness of Metacognitive Therapy (MCT) in the Treatment of Patients With Major Depressive Disorder (MDD)
Brief Title: Clinical Trial of the Effectiveness of Metacognitive Therapy in the Treatment of Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCTDEP
Record Dates: First submitted 2012-02-09; First posted 2012-05-31 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; psychotherapy; metacognitive therapy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive therapy (Experimental)
  Interventions: Behavioral: Metacognitive therapy
- Waiting list control (No Intervention)

INTERVENTIONS:
Behavioral: Metacognitive therapy — Metacognitive therapy, 10 weekly sessions of 45-60 minutes duration each
  Arms: Metacognitive therapy

SUMMARY:
The main aim of this study is to (1) evaluate the effectiveness of metacognitive therapy for major depressive disorder. Additional aims are to (2) investigate patterns of change and the mechanisms of action involved during treatment, and to (3) examine the impact of meta-cognitions in the treatment and relapse prevention of depression.

DETAILED DESCRIPTION:
Major depressive disorder is a disabling condition which adversely affects a person's family, work or school life, sleeping and eating habits, and general health.

Cognitive-behavioral therapy (CBT) is a recommended treatment for depression, with a large number of clinical trials supporting its efficacy. However, despite the success of CBT relative to other treatments, only 40-58 % of patients receiving CBT may be classified as recovered using clinical significant change assessed by the Beck Depression Inventory. Moreover, research demonstrates that only between one-third and one quarter of patients receiving CBT remain recovered at 18 months follow-up.

A new treatment approach to MDD is Meta-Cognitive Therapy. In this treatment approach, MDD is conceptualized as being maintained by rumination and meta-cognitions. Treatment seeks to challenge and change specific meta-cognitions and rumination, through behavioural experiments and verbal reattribution. No randomized controlled studies have compared the effectiveness of MCT to a waiting-list condition for MDD. Related to this, no study has examined the specific elements of therapy that are hypothesized to be of most importance for changing rumination, leading to positive treatment outcomes.

The purpose of this trial is to investigate the efficacy of Wells' MCT for Major Depressive Disorder (MDD). Another aim will be to examine the in-treatment processes associated with positive treatment outcomes.

The study will be a randomized controlled, trial comprising 50 patients with a primary diagnosis of major depressive disorder (DSM-IV; APA, 1994). Experienced diagnosticians will assess all patients by using structural interviews such as SCID-I, SCID II and the Hamilton Rating Scale for Depression.

All patients will be randomized in blocks to two groups in order to compare the following conditions: MCT and a wait list control condition. After the waiting period of 10 weeks, the patients in the wait-list condition will be allocated to the treatment condition. Both between-subjects and within-subjects comparisons will be conducted.

The research trial will be conducted at the outpatient-clinic at the Department of Psychology, Norwegian University of Science and Technology in Trondheim, Norway.

Questions that will be addressed:

1. Are the effects of MCT possible to replicate by a separate research group (other clinical groups than those that developed the method)?
2. Is MCT better than a waitlist condition?
3. Is change in positive and negative appraisals of rumination predictive of treatment outcome?
4. What is the effect size of MCT for depression? How is the relapse prevention of MCT?
5. Does the treatment have an effect on co-morbid anxiety disorder (s)?
6. What treatment elements predict outcome in MCT?
7. What effect does the treatment have on stable personality traits linked to depression and anxiety (e.g., neuroticism)?

The meta-cognitive treatment program is based on Wells' manual. The patients who are receiving meta-cognitive therapy will be treated up to maximum 10 sessions, with weekly session of 45-60 minute duration.

In the first treatment session, an idiosyncratic case formulation based on the MCT model of depression is built and shared with each patient. Socialization to the model then follows, which emphasizes how rumination and a high level of self focus (e.g., focusing on negative thoughts and feelings) maintains depression. At the end of the first treatment session, attention training (ATT) is introduced as a method of counteracting excessive self-focus, and to help patients' switch to a meta-cognitive mode of processing. ATT is an auditory attention task consisting of three stages; selective attention, attention switching and divided attention. The task takes approximately 10 minutes, and once practiced in session, patients are asked to implement ATT daily as a homework assignment. In-session practice of ATT is used throughout treatment.

In the next sessions, treatment focuses on a careful identification of rumination, and on modifying related positive and negative beliefs. Verbal reattribution strategies are used to modify negative beliefs concerning the uncontrollable nature of rumination. This is followed by training patients in 'detached mindfulness', coupled with rumination postponement experiments which challenge the belief that rumination is uncontrollable. Patients are asked whether they have ever noticed their negative thoughts, but chosen to not engage with them. In this context, engagement means rumination, analysis of the thought, cognitive avoidance or any form of further processing of the thought. Patients may still be motivated to use rumination as a coping strategy if positive beliefs about rumination remain. To counteract positive beliefs, an analysis of the advantages and disadvantages of rumination is undertaken to demonstrate that rumination maintains depression and is not an effective method of coping.

The final treatment sessions focused on relapse prevention and further modification of positive and negative meta-cognitive beliefs, including erroneous beliefs about the recurrence of emotion and deviations in mood. Relapse prevention further involves the development of a therapy blueprint which includes a written and diagrammatic formulation of the meta-cognitive model of depression. A detailed account of the main therapeutic strategies used during treatment is provided, along with a specific plan for the patient to implement in guiding their thinking and behavioral style in responses to future negative moods. Patients are encouraged to implement these strategies to maintain and strengthen the gains made over the course of treatment.

The treatment will be administered according to the originators published treatment protocols for MCT. Independent assessors will assess adherence and quality of treatment.

Independent experts will assess the quality of treatment by inspection of a sampling of video-recorded treatments. Using checklists session-by-session will ensure adherence of the therapy. Responsible investigator and supervisors will be using video of all treatment sessions to assess adherence to the treatment condition.

1. All patients referred to the university clinic will be consecutively assessed at intake (SCID-I + II, HDRS-17). Based on diagnosis and criteria for inclusion and exclusion, the patients will be asked to volunteer to participate in the study and confirm by signing a form of consent.
2. Patients will be randomized to one of two conditions.
3. Patients will be asked to self-rate symptoms on a battery of self-report questionnaires.
4. Meta-cognitive therapy will be given to patients in group 1, while group 2 is a waiting list control. Waiting list controls will be rated but not treated and will wait for treatment for 10 weeks.
5. After 10 weeks the waiting list controls will transferred to the treatment group.
6. The patients will be assessed prior to treatment, by 10 weeks in treatment, and at six months and at , one and two years of follow-up.
7. Reassessment of the diagnosis and symptom severity is made by post-treatment.

Criteria for recovery will be: Jacobsen criteria of a minimum change and patients crossing the cut-off point on two measures: The HDRS-17 and BDI. Other outcome measures will include:

* Reduction of depressive symptoms as measured by self-report questionnaires
* Number of patients with no MDD diagnosis based on SCID-I after treatment
* Relapse rate during six months and at , one and two years follow-up

The proportion of responders as measured by the HDRS-17 and BDI and those who no longer fulfil the conditions for a MDD diagnosis at post-treatment and by 6 months and one and two years follow-up.

The secondary efficacy variables will be the proportion of responders at post-treatment and six months and by , one and two years follow-up as measured by the other symptom measures. In addition, the proportions of responders as measured by MDD-S and the relapse rates during two one years of follow-up are selected to be one of the secondary efficacy variables.

A comparison between the two groups of patients will be conducted at post-treatment and there will be 6 month and at one- and two years of follow up for the treatment condition. The null hypothesis is assumed. A within group analyses will be conducted in order to estimate effect sizes and significant clinical change estimates.

Participants will be randomized in blocks of 17 patients divided on three conditions in a 1:2 ratio. Two factors are controlled for in the randomization. First, gender, second the number of previous depressive episodes (DSM-IV, APA 1994). A computer provided by NTNU will generate the randomization list.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder
* 18 years or older
* Signed written informed consent prior to entry in the study

Exclusion Criteria:

* Known somatic disease
* Psychosis
* Current suicide intent
* PTSD
* Cluster A or cluster B personality disorder
* Substance dependence
* Not willing to accept random allocation
* Not willing to withdraw psychotropic medication for a period of 4 weeks prior to entry to the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in depression | baseline (before treatment), week 1-11, 12 months follow-up
  Hamilton Depression Rating Scale (HDRS-17; Hamilton, 1967)
Change in diagnosis | baseline (before treatment), week 11, 12 months follow-up
  SCID I and II (First et al., 1995, 1997)

SECONDARY OUTCOMES:
Change in depression | baseline (before treatment), week 1-11, 6 and 12 months follow-up
  Major Depressive Disorder Scale (MDD-S; Wells, 2009)
Change in anxiety | baseline (before treatment), week 1-11, 6 and 12 months follow-up
  Beck Anxiety Inventory (BAI; Beck et al., 1988)
Change in automatic thought | baseline (before treatment), week 11, 6 and 12 months follow-up
  Automatic Thought Questionnaire (ATQ; hollon & Kendall,
Change in rumination | baseline (before treatment), week 11, 6 and 12 months follow-up
  Rumination Response Scale (RRS; Nolen-Hoeksema & Morrow, 1991)
Change in positive beliefs | baseline (before treatment), week 11, 6 and 12 months follow-up
  Positive beliefs about Rumination (PBRS; Papageorgiou & Wells, 2001)
Change in negative beliefs | baseline (before treatment), week 11, 6 and 12 months follow-up
  Negative Beliefs about Rumination (NBRS; Papageorgiou & Wells, 2008)
Change in metacognitions | baseline (before treatment), week 11, 6 and 12 months follow-up
  Metacognitions Questionnaire-30 (MCQ-30; Wells & Cartwright-Hatton, 2003)
Change in resilience | baseline (before treatment), week 11, 6 and 12 months follow-up
  Resilience Scale for Adults (RSA; Friborg & Hjemdal, 2003)
Change in interpersonal problems | baseline (before treatment), week 11, 6 and 12 months follow-up
  Inventory of Interpersonal Problems (IIP-64; Horowitz et al., 1988)
Change in worry | baseline (before treatment), week 11, 6 and 12 months follow-up
  Penn Scale Worry Questionnaire (PSWQ; Meyer et al., 1990)
Quality of working alliance | week 3
  Working Alliance Inventory (Horvath & Greenberg, 1989)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hagen, PhD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of psychology, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Background] Hjemdal O, Solem S, Hagen R, Kennair LEO, Nordahl HM, Wells A. A Randomized Controlled Trial of Metacognitive Therapy for Depression: Analysis of 1-Year Follow-Up. Front Psychol. 2019 Aug 8;10:1842. doi: 10.3389/fpsyg.2019.01842. eCollection 2019. PMID 31440193
- [Result] Hagen R, Hjemdal O, Solem S, Kennair LE, Nordahl HM, Fisher P, Wells A. Metacognitive Therapy for Depression in Adults: A Waiting List Randomized Controlled Trial with Six Months Follow-Up. Front Psychol. 2017 Jan 24;8:31. doi: 10.3389/fpsyg.2017.00031. eCollection 2017. PMID 28174547